CLINICAL TRIAL: NCT00752245
Title: Study of the Kinetics of Uremic Toxins in the ICU Patients With Acute Renal Failure, in Order to Optimize the Dialysis Dose: Patients With Sepsis/Multi-organ Failure
Brief Title: Uremic Toxins in the Intensive Care Unit (ICU): Patients With Sepsis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008/373
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Renal Failure; Multi Organ Failure
Keywords: ICU patients with acute renal failure with sepsis/multi-organ failure
MeSH Terms: conditions — Renal Insufficiency; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Dialysis during 4 hours
  Interventions: Procedure: Dialysis during 4 hours
- 2 (Active Comparator): Dialysis during 6 hours
  Interventions: Procedure: Dialysis during 6 hours
- 3 (Active Comparator): Dialysis during 8 hours
  Interventions: Procedure: Dialysis during 8 hours

INTERVENTIONS:
Procedure: Dialysis during 4 hours — Blood and dialysate sampling
  Arms: 1
Procedure: Dialysis during 6 hours — Blood and dialysate sampling
  Arms: 2
Procedure: Dialysis during 8 hours — Blood and dialysate sampling
  Arms: 3

SUMMARY:
Study of the kinetics of uremic toxins in the ICU patients with acute renal failure, in order to optimize the dialysis dose: patients with sepsis/multi-organ failure. The sampling of blood and dialysate will be done during dialyses with different durations (4, 6 and 8h)

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with sepsis/multi-organ failure with acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07-31 (Actual); Primary Completion 2013-10-04 (Actual); Study Completion 2013-10-04 (Actual)

PRIMARY OUTCOMES:
Registration of toxin removal efficiency | During dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be